# INFORMED CONSENT TO TAKE PART IN A CLINICAL RESEARCH STUDY AND AUTHORIZATION TO USE AND DISCLOSE MEDICAL INFORMATION

**TITLE:** A Phase 1, Randomized, Double-Blind, Placebo-Controlled,

Dose-Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Intravenous Ertapenem in Combination with

Zidebactam (WCK 6777) in Healthy Adult Subjects

PROTOCOL NO.: DMID 21-0013

**PURPOSE:** Multiple drug-resistant infection

**TYPE OF STUDY:** Phase I – HEALTHY SUBJECTS

**SPONSOR:** Division of Microbiology and Infectious Diseases (DMID)

National Institute of Allergy and Infectious Diseases (NIAID)

National Institutes of Health (NIH) 5601 Fishers Lane, MSC 9806 Bethesda, Maryland 20892

**STUDY DOCTOR:** Martin Kankam, MD, PhD, MPH, FAPCR

**RESEARCH SITE** Altasciences Clinical Kansas, Inc.

ADDRESS: 10103 and/or 10203 and/or 10183 Metcalf Avenue

Overland Park, KS 66212

**TELEPHONE NUMBER** 913-696-1601 (24-hour number)

#### **KEY INFORMATION**

The following is a summary of the things you should know about this clinical research study:

• You are invited to take part in a clinical research study of the drugs ertapenem (ERT) and zidebactam (ZID), which will be administered separately, or combined (ERT-ZID or WCK 6777). This means that the study drugs are allowed to be evaluated in healthy persons like you in this study by the U.S. Food and Drug Administration (FDA), but not approved for use in people by prescription. Your participation is voluntary and your consent to participate is sought after you have read and understood information provided in this document and have your questions about the study answered before any study tests are done. If you consented and then change your mind, you may withdraw from the study and notify the study doctor. If you withdraw after you received even a dose of a study drug, you will have a medical evaluation and lab tests to ensure you are doing well and you will be asked to consent to remain in the study for more safety follow up and possibly for some more blood sampling for measuring the study drug concentration in your blood.

- Zidebactam (ZID) is a compound that is being developed for use in combination with other antibiotics, such as with ertapenem (ERT), for the treatment of severe infections that are resistant to multiple available antibiotics. Ertapenem (ERT) is an antibiotic approved by the FDA for use in people for the treatment of various infections. In this study, ERT will be used in doses higher than approved by the FDA. In this study, ZID and ERT will be studied alone and in combination. The combination of ERT and ZID is called WCK 6777 and will be used in people for the first time in this study.
- The purpose of this research study is to collect information about the safety of taking ZID and ERT alone or in combination (WCK 6777), that is, if any side-effects occur after taking them, and their type and how severe they are. Information will also be collected about the study drug pharmacokinetics (PK), that is, how the body handles the drugs after taking them at the doses to be used.
- You will be assigned to one of 7 study treatment cohorts (groups), numbered 1 to 7. Some cohorts will have both study drugs (Cohorts 1, 4 and 7) and others only ERT (Cohort 2 and Cohort 5) or only ZID (Cohort 3 and Cohort 6). The cohorts will run sequentially in the order they are numbered, that is, Cohort 1 will be done before Cohort 2, etc. and the lowest dose will be in Cohort 1 and the highest in Cohort 7.
- A total of 52 subjects will take part in the study, 8 subjects each in Cohorts 1, 2, 4, 5, and 7 and 6 subjects each in Cohorts 3 and 6. In Cohorts 1, 2, 4, 5 and 7, you will be assigned randomly (like tossing a coin) to receive either the study drug (75% chance) or placebo (saline, salt water) (25% chance). In Cohorts 3 and 6, you will receive only the designated study drug.
- The study drug(s) or placebo will be infused intravenously (IV; in a vein) once a day for 7 days, and the volume and duration of each infusion will vary depending on the cohort you will be assigned to: 100 mL (about 3.5 ounces) over 30 minutes in Cohort 1, 250 mL (about 8.5 ounces) over 60 minutes in Cohorts 2, 3 and 4 and 250 mL (about 8.5 ounces) over 120 minutes in Cohorts 5, 6 and 7.
- If you decide to participate, you will be in the study for up to 42 days (from Screening Visit to Final Visit). There is a *Screening Period* of up to 27 days to determine if you meet the study requirements; an *Inpatient Period* of 9 days/8 nights, with 1 day to check-in, to confirm you can take part in study and be admitted in the clinical research site, 7 days with daily dosing with the study drug or placebo assigned to your cohort, and 1 day of evaluations before discharge; and an *Out-patient Follow-up Period* with one final visit to the research site between 4 to 7 days after receiving the last dose of the study drug.
- Screening evaluations will start after signing this form to document your willingness to take part in this study. We will collect demographic information about you (age, sex, race and ethnicity) and social habits (smoking, alcohol use, drug use, exercise). Medical evaluations will include your medical and surgical history, history of medications you take, physical examination (PE), measurement of your body weight and height, taking your vital signs (VS;

measurement of blood pressure, heart rate, breathing rate and temperature), blood and urine tests, test for hepatitis and HIV, a pregnancy test if you are female, a test to confirm if you are postmenopausal if you are female, and an electrocardiogram (ECG; paper tracing of the heart signals). If you meet all the requirements to take part in the study, you will be given an appointment to check-in in the clinical research site 1 day before starting study drug administration to confirm that you continue meeting the requirements to participate in the study.

- Starting on Day 1 and until Day 7, you will receive a single IV dose of the study drug or placebo according to the cohort (group) you are in. The effects of the study drug on you will be assessed by your reports of symptoms and responses to questions by the clinical staff, physical exams focused on the symptoms you have, vital signs, and blood and urine laboratory tests at various timepoints after you received the study drug and until your last visit. Blood and urine samples will also be collected during these days to measure the drug concentration and study the drug pharmacokinetics (PK, how your body handles the drug). Blood will be drawn from a vein in the arm opposite the one for infusion. You will be discharged from the clinical site on Day 8 and return to the clinical site between Day 11 and 14 for your final out-patient visit.
- Risks that could be caused by the study drugs are:
  - O Zidebactam (ZID) was safe and well-tolerated in previous studies in healthy people in doses the same or higher than the doses to be used in this study. The most common side effects thought to be related to the study drug were:
    - Mild to moderate headache
    - Injection site irritation (pain, redness)
  - Zidebactam's potential to cause mutations and cancer needs further testing, and there are no long-term studies to evaluate this risk in animals and humans. However, this risk is considered low because the study drug will be administered only up to 7 times (doses) in this study.
  - o Ertapenem (ERT) was safe and well-tolerated as a standalone drug by patients at the FDA approved dose (1 gram daily) after it was approved as a prescription drug. In this study, ERT will be used at higher doses than the approved dose, and these doses (2 grams and 3 grams daily) were found to be safe and well-tolerated in research studies in healthy people. The most common side effects thought to be related to the drug were:
    - Mild to moderate diarrhea
    - Nausea
    - Vomiting
    - Headache
    - Somnolence (increased tendency to sleep)
    - Dizziness
    - Vein irritation at the infusion site
    - Vaginitis in females
    - Increase of liver enzymes
    - Increase of platelet counts in the blood

- o Potential side-effects of ertapenem are:
  - An allergic reaction
  - Muscle tremor
  - In the higher doses (2 grams and 3 grams) that will be used in this study, the following may occur:
    - Nausea
    - Diarrhea
    - Brief dizziness
- o WCT 6777 (ERT+ZID combination) has not been studied before in people. Side effects could be those of each of the study drug components or others that are not known.
- Risks that could be caused by the study procedures are:
  - o There may be side effects of inserting needles or a catheter in the vein to collect blood or for an IV infusion. Local pain, bruising, bleeding, phlebitis (inflammation or infection of the vein) or thrombophlebitis (clotting of blood in the vein) might occur at the site of the needle stick or IV catheter. There is a possibility of dizziness or fainting while your blood is being drawn.
  - There may be side effects of blood draws, such as dizziness standing or feeling tired, which may be caused by decreased blood volume or anemia (low blood counts). The amount of blood that will be drawn is less than the volume drawn in a blood donation.
  - There could be side effects from the ECG patches, such as a rash or minor irritation of the skin with itching. There could also be a need to shave a small area of the skin to place the patch.
- The study staff will monitor your well-being during the study, evaluate you medically, and provide appropriate treatment as required. Precautions will be taken to minimize complications from blood draws or IV infusions.
- The study has no direct benefit for you. Knowledge gained in the study could be of future benefit to public health and to individuals with infections, who might benefit if the study drug is licensed. You will be promptly notified of any abnormal clinical test results that may suggest previously unknown abnormalities that could be clinically significant, and you will be counseled to see your own doctor for follow up.
- There are no alternatives to the research study. You are free to consent to participate in the study or not to participate or to withdraw after you consented initially. You will be compensated for the study days and procedures you complete. You will not be penalized if you withdraw from the study.
- Your personal health information will be protected. Your study medical record, laboratory test results and storage tubes containing your blood (plasma) and urine specimens will be coded and will not identify you by name or provide any other personal information that can identify you.

#### INTRODUCTION

You are being asked to be a volunteer in a clinical research study. You cannot be in this study if you are in another research study or have been in another study within the past month. Before you agree to be a part of this study, it is very important that you read and understand the study plan and in what ways you will need to cooperate. This consent form may have words in it that you do not understand. You may ask the study doctor or the study staff to explain any words or information that you do not understand. If you sign and date this form, it means you want to be in this study.

This form describes the reason for the study, and the way the study will be done. It also describes the benefits, risks, discomforts, and warnings about the study. This form will also explain how your medical information will be used, and who may see it. It describes your rights as a volunteer in the study.

The study staff will ask you many questions. Your answers must be completely truthful. Your health history and any changes in the way you feel during the study are very important. You must tell the study staff about any changes in your health or the way you feel. If you are not truthful, you may harm yourself by being in this study. Your signature on this consent form serves as proof of your promise that the information you give is true and correct and that you will remain truthful during this research study.

Altasciences Clinical Kansas, Inc., the research site, is being paid by the Division of Microbiology and Infectious Diseases (DMID) of the National Institute of Allergy and Infectious Diseases (NIAID), part of the National Institutes of Health (NIH). DMID is also referred to as the "study sponsor" in this document.

# **BACKGROUND AND PURPOSE**

The study doctor and the Division of Microbiology and Infectious Diseases (DMID) and the drug company, Wockhardt, Ltd, are conducting this research study of WCK 6777 (ZID-ERT), an investigational combination of two study drugs, Zidebactam (ZID) and Ertapenem (ERT). Zidebactam (ZID) is an investigational drug that has been allowed by the Food and Drug Administration (FDA) to be used in humans in research studies only. Ertapenem (ERT) is an antibiotic approved by the FDA for human use in 2001. The doses of ERT to be used in this research study are higher than the max daily dose recommended by prescription. This research study is the first one where the combination of ZID with ERT, called WCT 6777, will be studied.

**ZID** is a synthetic antibiotic that was made to combat infections against bacteria that are resistant to existing antibiotics. It can block some bacterial proteins that cause resistance to available antibiotics and enhances (boosts, makes stronger) the effect of other antibiotics, like ERT, to which bacteria are developing resistance. In animals, ZID increased the ability of other antibiotics to kill of some of the most resistant bacteria known that are the cause of severe kidney, lung and abdominal infections in people. ZID in combination with another antibiotic called cefepime is in advance testing for the treatment of urinary (kidney) infections in people. In this study, ZID will be evaluated in combination with ERT.

**ERT** is a synthetic antibiotic that has been approved by the Food and Drug Administration (FDA) and has been used extensively in the last 21 years for the treatment of severe skin, kidney, lung, abdominal and other infections in people from age 3 months and up. ERT is considered investigational in this study because it will be used in doses higher than recommended by prescription. It is also studied in combination with ZID because it was found that bacteria that were no longer sensitive to ERT or to ZID alone in the laboratory were sensitive to the combination of the two study drugs.

WCK 6777 (ERT+ZID) is a combination of these two antibiotics, ERT and ZID, that has shown to be effective against resistant bacteria in the lab and in animal studies. The combination is evaluated in healthy persons before it is tested in people with infections in order to understand the safety profile and the PK of the two antibiotics used together. It is expected that the combination will be effective in infections for which the number of existing effective antibiotics becomes smaller. The combination of the two study drugs could also be given in an outpatient facility as an IV infusion that is completed in relatively short time, something that could cut down hospitalization time and cost.

This research study will evaluate the effects of progressively increasing doses of either ZID or ERT alone or WCK 6777 (ERT+ZID combination) when administered IV as single daily doses for 7 days. The overall goals are to determine the safety, tolerability, and pharmacokinetics (PK) of the study drugs and if there are interactions when given together. Pharmacokinetics is the study of how a drug is absorbed, distributed, metabolized, and eventually eliminated by the body.

This study will be conducted in adults between 18 to 45 years of age who are in good health, do not take certain medications, and, for women, if they are not pregnant or breastfeeding. There will be a total of approximately 52 male and female subjects in this study. This study will be done at one site in the United States. All subjects in this study will receive a single IV dose of either the study drug or the combination of the two study drugs daily for 7 days.

The study will take up to 42 days to complete and is made up of the following periods: a *Screening Period* up to 27 days (Day -28 to Day -2), during which you will have screening tests if you consent to participate; a *Check-in* day (Day -1) to confirm your eligibility and, if you still qualify, to admit you in the research site and enroll you in the study; an *Inpatient Study Treatment Period* lasting 9 days/8 nights, with eligibility reviewed prior to study treatment administered on Day 1, and once daily doses of the study drugs or placebo from Day 1 to Day 7, and discharge from the Research Site on Day 8; and an *Outpatient Follow-up Period* of up to 6 days, with a single, last visit to the Research Site on Day 11 (+3 days) (4 to 7 days after the last study treatment).

A description of this research study will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the study results. You can search this website at any time.

# INFORMATION ABOUT THE STUDY

If you are eligible to take part in this study, you will receive either one of the study drugs or their combination according to the cohort (group) you were screened for. The study drug(s), doses of each drug, and the volume and duration of infusion in each cohort vary and are as follows:

| COHORT | STUDY | STUDY<br>DRUG DOGE | INFUSION VOLUME | INFUSION |
|---|---|---|---|---|
| NUMBER | DRUG | DRUG DOSE | | DURATION |
| 1 | WCK 6777 | 1 gram ERT | 100 mL (about 3.5 ounces) | 30 minutes |
| | or placebo | + 1 gram ZID | 100 IIIL (about 3.5 ounces) | |
| 2 | ERT | 2 grams ERT | 250 mL (about 8.5 ounces) | 1 hour |
| | or placebo | 2 grains EK1 | 230 IIIL (about 8.3 ounces) | |
| 3 | ZID | 2 grams ZID | 250 mL (about 8.5 ounces | 1 hour |
| 4 | WCK 6777 | 2 grams ERT | | 1 hour |
| | or placebo | + 2 grams ZID | | 1 nour |
| 5 | ERT | 2 ~~~ EDT | 250 m.L (about 9.5 ann acc | 2 hours |
| | or placebo | 3 grams ERT | 250 mL (about 8.5 ounces | |
| 6 | ZID | 3 grams ZID | 250 mL (about 8.5 ounces | 2 hours |
| 7 | WCK 6777 | 3 grams ERT | 250 mL (about 8.5 avecas | 2 hours |
| | or placebo | + 3 grams ZID | 250 mL (about 8.5 ounces | 2 nours |

Each subject in each cohort, except Cohort 3 and Cohort 6, will be randomized (like tossing a coin) to receive either study drug or placebo (salt water for infusion). The chance of receiving placebo is 25%. Additional subjects may also be admitted to the Research Site before dosing and may serve as back-up study subjects. You may be selected to participate in this research study as either a study subject or a back-up study subject. If you were selected as a back-up but did not receive a study treatment, you could be placed in the same cohort or another one if you are still interested in taking part in the study.

On Days 1 to 7, you will have a catheter inserted into a vein in the hand or arm for taking blood and another catheter for infusing the study drug or study drug combination in the opposite arm. The infusion volume and duration of infusion will vary depending on the cohort you are in: For Cohort 1, the volume will be 100 mL (about 3.5 ounces) and the infusion will last 0.5 hours (30 minutes); for Cohorts 2, 3 and 4, the volume will be 250 mL (about 8.5 ounces) and the infusion will last 1 hour (60 minutes); and for Cohorts 5, 6 and 7, the volume will be 250 mL (about 8.5 ounces) and the infusion will last 2 hours (120 minutes). After dosing with study drug, you will be monitored daily, and data will be collected to evaluate the effect of the study drug on you. After the dose on Day 1, you will have frequent blood samples taken for the next 24 hours to measure the concentration of study drug in the blood, and you will be asked to collect all your urine samples during the same period. Blood and urine collections up to 24 hours after the dose will also be done on Day 7.

You will be asked to come to the Research Site 3 times: 2 times before receiving the study drug, and 1 time after receiving it. You will be admitted in the Research Site on Day -1 after you complete testing on the second visit and stay in the Altasciences Clinical Kansas research site for 8 nights/9 days if you meet the requirements for receiving the study drug.

The first visit will be a **screening visit**. You will be informed about the study, have your questions answered and, if you decide to participate in the study, as shown by signing and dating this consent form, you can proceed to the first part of screening to evaluate your eligibility to take part in the study. If you decide to participate and sign this consent form, we will collect your demographic information (age, sex, race, ethnicity) and social habits (smoking, alcohol and drug use, exercise), The medical evaluations will include your medical and surgical history, history of prescription and non-prescription medications you take, a physical exam (PE), measurements of your height and weight and of your vital signs (VS; blood pressure, heart rate, breathing rate, and temperature), an ECG (a paper tracing of your heart beats), standard blood tests (blood counts, chemistries, coagulation tests) and urine lab tests, a pregnancy test if you are female, a test to confirm if you are post-menopausal if you're female, tests for hepatitis B and C and for HIV, and urine tests for drugs, alcohol, and cotinine.

If you pass the screening tests, you will be asked to return to the Research Site for a second visit on (**Day -1, Check-in**) to complete medical and lab tests and confirm that you can be admitted. If you continue to be eligible to continue participating in the study, then you will stay in the Research Site overnight for the inpatient study treatment period.

o If you do not pass the screening test, the study staff will tell you why and may counsel you to seek medical attention based on any abnormal lab tests or other findings.

On the next day (**Day 1**), you will begin the **inpatient study treatment period** of the study. In the morning on Day 1, you will have baseline VS and collection of plasma and urine for PK. You will be required to have no food to eat for at least 4 hours before the IV study treatment infusion. Catheters will be inserted in a vein in one arm to infuse the study drug and in another vein in the other arm to draw blood. You will receive the study drug or placebo IV through the vein, The volume and duration of duration of infusion will vary depending on the cohort you are in (see the table on page 6). You may eat food 1 hour after the end of the infusion. In the next 24 hours, you will have 7-9 blood draws at scheduled times, each about 2 teaspoons, to measure the study drug concentration in the blood (plasma PK). You will also start collecting all the urine at intervals for the measurement of the study drug (urine PK) until 24 hours after the start of dosing. The last PK will be completed before you receive the next dose of study drug on Day 2.

# Recording and evaluating side-effects will start with the first dose and continue through the end of the study.

On **Days 2 to 6**, you will have an IV infusion of the study drug daily, in the same volume, study drug dose, for the same duration and starting about the same time as on Day 1. You may eat food 1 hour after the end of the IV infusion. You will have vital signs taken before infusion. You will have blood drawn for lab tests before dosing on Days 2, 4 and 6. Plasma PK blood draws will be collected before each dose on Days 2, 3, 4, 5 and 6 and 12 hours after the dose. The catheters in your veins may stay in up to 3-4 days, but they may be removed more frequently if your veins are irritated or the catheters do not work, and new catheters will be placed in your veins.

On **Day 7**, you will have the last dose of study drug or placebo infused IV as on Day 1. You will have medical assessments Plasma and urine PK will be collected at scheduled times for 24 hours after the study drug infusion, until the morning of Day 8, exactly as it was done on Day 1.

On **Day 8**, you will complete required medical and lab testing. You will be counseled to avoid prohibited drugs, avoid pregnancy and continue contraception for 30 days after last dose of the study drug. If you are a male, you will be counseled not to donate sperm for 30 days after the last dose of study drug and, for you and your partner to use appropriate contraception for the same period. Then you will be discharged from the research site after you complete all your evaluations.

On **Day 11 (+3 days)**, that is 11 to 14 days after the first dose (4 to 7 days after the last dose), you will be asked to return to the research site to complete required final medical and lab evaluations.

You will be asked for any new symptoms before the first dose and continue until you complete the study on the last visit. You will have additional physical exams and lab tests as needed for the evaluation of any new symptoms and findings that you may have. You may be asked to return to the research unit to follow up on any abnormal lab tests or other findings as necessary until they are no longer present, or they are not clinically significant in the judgement of study doctors.

The schedule for screening, check-in / enrollment study treatment, and outpatient follow-up periods is shown in the table below:

| Outpatient<br>Screening | Inpatient | Inpatient Study<br>Treatment | | Outpatient<br>Follow Up |
|---|---|---|---|---|
| Screening Period | Check-in/<br>Enrollment | Dosing | Discharge | Final Visit |
| Day -28 to Day -2 | Day -1 | Day 1 to Day 7 | Day 8 | Day 11 (+3 days) |

#### **MEDICAL MONITORING**

The study staff will monitor you for side effects during your stay in the Research Site and provide medical care as needed if you have any medical problems. Guidelines have been created to evaluate the safety of the study drug. If you have any side effects, we will evaluate your symptoms and treat you as indicated according to standard medical practices.

# WHAT WILL HAPPEN DURING THE STUDY?

#### SCREENING PERIOD (Day -28 to Day -2)

# **SCREENING VISIT:**

During this visit, you will be informed about the study, have your questions answered and, if you decide you want to participate in the study, show your intent by signing and dating this consent form.

After signing this consent and before you begin the study, you will have the following screening tests done to determine if you are in good health and qualify to continue participation in the study:

- Complete medical history (including your demographic information) and medication review.
- Vital signs (VS; blood pressure, heart rate, breathing rate and oral temperature) and height and weight measured, and Body Mass Index (BMI) calculated.
- Complete a Physical Examination.
- Have a 12-lead ECG (standard recording) This will require attachment of electrodes from the standard ECG machine to your chest, arms, and legs. Male subjects may have to have their chest hair shaved for the ECG. Female subjects may not be allowed to wear a bra during ECG-related procedures.
- You will have blood and urine collected for laboratory tests (you will be asked to not eat or drink anything other than water for at least 4 hours before blood collection).
- You will have a urine test for alcohol, and urine drug screen for illegal drugs and cotinine (for detecting nicotine products). (The tests must be negative to qualify.)
- Blood collected for serum pregnancy test if female. (The test must be negative to qualify.)
- Blood collected for measurement of follicle-stimulating hormone (FSH) if post-menopausal female.
- Testing for Hepatitis B, Hepatitis C, and HIV infections: Your blood will be tested for the HIV antibody. HIV is a virus that causes AIDS. You will also be tested for Hepatitis B and C Viruses. (Test results must be negative to qualify.)
  - Note that it may take weeks or months after being infected with HIV for the test to be positive. If you have a positive HIV or hepatitis test, you cannot be in the study. If the HIV or hepatitis test are positive, you will be notified by the Research Site and given information on how to follow up for further medical care. As required by law, positive test results must be reported by the Research Site to the State Department of Health. If you have any questions about what information is required to be reported, please ask the study staff. If the Research Site becomes aware during your participation in this study that there is any change in the HIV or Hepatitis Virus results, you will be withdrawn from the study. Your test results are private (confidential); however, this cannot be guaranteed. For example, it is possible for a court of law to get health or study records without your permission.

You will be told of the results of medical tests and whether you can continue participating in the study.

- If you do not meet the study requirements, you will be discharged from the study. You will be told why you were not selected for the study.
  - o If there is a medical condition or abnormal laboratory test that needs further medical attention, you will be counselled to follow up with your primary doctor or contact community physicians or clinics where you can go for testing and follow up. You may sign a release form to allow the Research Site to release medical tests to you or send them to your own doctor or clinic.
- If your medical tests are good and confirm your eligibility to participate in the research study, the study staff will ask you to return to the Research Site on Day -1 to complete the inpatient screening tests to confirm your eligibility to participate in the study.

- You will be told to come prepared to stay for the inpatient study treatment if you pass the tests.
- You will be counselled to avoid pregnancy, use appropriate contraception (both male and female), and avoid prohibited medications, tobacco and other nicotine products, alcohol, and marijuana and illegal drugs.
- o You should avoid strenuous physical activity.

# CHECK-IN VISIT (Day -1) (1 day before the study treatment period)

On this day, you will have the same tests as you did at the Screening visit to confirm that you continue being in good health and meet the requirements for admission and receiving the study drugs. The study doctor will review the results of your tests to see if you still qualify.

- If you do not meet the study requirements, you will be discharged on this day. You will be told why you were not selected for the study. If there is a medical condition or abnormal laboratory test that needs further medical attention, you will be counselled to follow up with your primary doctor or contact community physicians or clinics where you can go for testing and follow up. You may sign a release form to allow the Research Site to release medical tests to you or send them to your own doctor or clinic.
- If you meet the study requirements, you will be admitted to the Research Site.

After you are admitted, you will complete an orientation of the in-patient facility, and asked to read the House Rules that describe what you are expected to follow while you stay in this facility and participate in the study.

- You will be told what study treatment cohort you were assigned to and review the procedures that will be performed during the Inpatient Study Treatment period. You will not be told if you are going to receive active study drug or placebo if you are assigned to a cohort where either one will be used (Cohorts 1, 2, 4, 5, and 7).
- You will be counseled to avoid excessive exercise.
- You will be encouraged to drink plenty of fluids to keep well hydrated.
- You will receive dinner and snacks in the Research Site.
- You will not be allowed to eat anything for 4 hours before taking the study drug the following morning, but you will be allowed to drink water during that period.

# **INPATIENT STUDY TREATMENT PERIOD (Days 1 to 8)**

You will receive the study drug daily in the morning on Days 1 to Day 7 and followed as inpatient until Day 8. The following procedures will be done during this period:

# **DAY 1 and DAY 7 (In-patient Dosing):**

#### Before Dosing:

• You will not eat any food or drink (other than water) at least 4 hours before taking the study drug (dosing). That means that you may have an evening snack the night before dosing but no food afterwards, and you will not eat breakfast before dosing. You will be allowed to drink water during that time before dosing.

- If you have new symptoms, you will have a physical exam and any medications you took will be reviewed and your vital signs measured. The results of the above will be reviewed to see if you still qualify to receive the study drug.
- You will have an IV catheter placed in a vein in your forearm to infuse study drug. You will have another IV catheter placed in a vein in your other arm to draw blood.
- You will have blood (plasma) PK and urine PK samples collected for analysis of study drug before dosing starts.
- You will be asked to empty the bladder as close to the start of the study drug infusion as possible.
- You will be encouraged to keep well hydrated starting before the study drug infusion and continue until 24 hours after the last dose.

#### Dosing:

• You will receive the study drug or placebo by IV infusion (in a vein) using an infusion pump in a volume and duration of infusion specified for the study drug or study drug combination selected for your cohort (See the table on page 6).

#### After Dosing Starts:

- You should report any side effects that you may experience after infusion starts until the end of the study. You will also be observed for side-effects during the infusion.
- You will have a physical exam done as needed for evaluation of new symptoms after dosing starts until the end of the study.
- Any medication that you take will be recorded to the end of the study.
- You will not eat solid food during the infusion and at least 1 hour after the end of the infusion but be able to drink water and non-carbonated beverages.
- You will have your vital signs measured.
- You will have blood drawn to measure the concentration of study drug approximately 7-9 times after you started receiving the study drug, depending on the cohort (group) you were assigned to.
- You will be asked to collect all urine for the next 24 hours in pools every 4 hours as follows: from the start of dosing to 4 hours, 4-8 hours, 8-12 hours, and 12-24 hours. Study staff will instruct you on how to collect the urine at various intervals.
- You will have the infusion site and the blood drawing site checked periodically by the study staff. Let the study staff know if you experience any discomfort or other symptoms at these sites.
- The study staff will let you know if they will keep the IV infusion line and blood draw line open to be used on the following day or removed and replaced.
- You may be served a meal 1 hour after the infusion. Let the study staff know if you have any nausea and you cannot eat.
- You will be encouraged to keep well hydrated.
- You will be counseled to avoid excessive exercise until the study end.

# DAY 2 to DAY 6 (In-patient Dosing):

### Before Dosing:

- You should report any side effects that you may experience.
- Any medication that you take will be recorded to the end of the study.
- Your infusion site and blood draw line will be examined, and new catheters inserted if needed.
- Your vital signs will be measured.
- You will have blood samples collected for clinical lab tests (Days 2, 4 and 6 only).
- You will have blood (plasma) drawn to measure the concentration of study drug daily within 30 min before dosing.
- You will be asked to finish the collection of urine for measuring the concentration of study drug within 30 min before dosing (Day 2 only).

# Dosing:

• You will have the study drug or placebo infused IV (in a vein) as on Day 1.

## After Dosing Starts:

- You should report any side effects that you may experience after infusion on each day.
- You will be observed for side-effects during the infusion.
- You will have a physical exam for evaluation of your symptoms.
- Any medication that you take will be recorded to the end of the study.
- You will have assessments after dosing on those days that are identical to those done on Day 1.
- Your study drug infusion IV line will be removed.
- You should continue good hydration daily.
- You will be counseled to avoid excessive exercise.

### **DAY 8 (Inpatient Follow-up):**

- You should report any side effects that you may experience. after infusion starts until the end of the study.
- You will have vital signs and weight measured, and an ECG recorded.
- You will have blood and urine samples collected for clinical laboratory tests.
- You will have blood (plasma) drawn to measure the concentration of study drug at 24 hours after last dose on Day 7.
- You will complete the collection of urine to measure the concentration of study drug at 12-24 hours after last dose on Day 7.
- You will have the IV infusion site examined and the IV blood draw catheter removed. You should report any discomfort you have at the infusion or blood draw site.
- You will have a complete physical examination.
- You will be discharged from the Research Site after review of clinical laboratory tests, ECGs, and other assessments by authorized clinician.

- You will be counseled to avoid pregnancy, continue contraception for 30 days after the last dose, avoid donating sperm for 30 days after last dose if you are a male, and avoid excessive exercise.
- You will be provided contact information and instructions to report to the Research Site any side effects or new symptoms that you develop during these periods and any medication that you take.
- You will be given an appointment to return to the Research Site to have follow-up tests on Day 11 (+3 days) after first dose (4 to 7 days after last dose).

# DAY 11 (+3 days) (Out-patient Follow-up – Final Visit):

- You should report any side effects that you may have experienced after your discharge from the research site on Day 8.
- You will be asked to report any medications that you took after your discharge from the research site on Day 8.
- You will have vital signs measured, and an ECG recorded
- You will have blood and urine samples collected for clinical laboratory tests.
- Your IV infusion site and IV blood draw site will be examined. Report any discomfort you have at the infusion or blood draw site.
- You will have a complete physical examination
- You will be counseled to avoid pregnancy, continue contraception for 30 days after the last dose, if you are a male avoid donating sperm for 30 days after last dose, and avoid excessive exercise.
- You should report any side effects that you may experience. You may be asked to return for an unscheduled visit for any symptoms that you may have.

The study staff will notify you if you have completed the study or if you must return to the research site for any lab tests that need be followed.

#### **EARLY TERMINATION:**

If you choose to withdraw from the study or are terminated by the investigator before you complete the study, you may be asked to consent to remain in the study to complete safety and PK blood collections. If you do not consent to remain in the study, you will have the same tests and procedures as described for Day 11 (Final Visit).

# **UNSCHEDULED VISIT (if needed):**

You may return to the Research Site for an unscheduled visit at any time after your discharge on Day 8 or after the last visit (Day 11) if you have any symptoms that you want to discuss or because the study staff asked you to come in for an evaluation. The following activities could be done according to the reason of your extra visit:

- You will be asked to provide information on the side-effects you may experience.
- You will be asked to document medications you take.
- You may have the Vital Signs measured.
- You may have a physical examination.
- You may have a 12-lead ECG if needed.

- You may have blood drawn and/or urine collected for clinical laboratory tests, if applicable.
- The study staff will give you information and tell you if you need to return for follow up for another visit.

The study staff may also request to have procedures performed that are not listed above to ensure your safety throughout the study.

# ADDITIONAL DRUG AND ALCOHOL SCREENS

Random urine drug and alcohol screens may be repeated at any time during the study if the study staff suspects alcohol or drug use. If you test positive for drug or alcohol use at any time after the first dose of study drug, you may be discontinued from the study.

#### CONTROLLED SEARCH

Designated study staff reserves the right to do a controlled search by having you put on a gown in order to have your clothes and person checked for disallowed items that may have been brought into the research site. This search involves removing all undergarments as well as putting on a gown so that there is no place the disallowed items could be kept.

At each admission into the research site, a search of your clothing, like pockets, and bags will occur. You will not be required to remove your clothing or undergarments, but staff may ask you to turn your pockets inside out or check areas of clothing that could conceal restricted items. Study staff will also perform a bag check and confiscate any items not permitted to be brought into the research site. These belongings will be returned to you at discharge from the research site.

#### **BLOOD SAMPLES**

Blood samples will be drawn by single needle-sticks or through an IV catheter, as determined by the study staff. An IV catheter is a small plastic tube inserted into your arm vein by a needle. The needle is removed, but the tube temporarily remains in your vein. This tube allows the removal of blood without having to stick you each time. It will be removed every 3-4 days or sooner if not working well or if you have local pain or vein irritation. The total amount of blood drawn will be up to about 371 mL (about 12.5 oz, a bit over a cup) during the in-patient study treatment period (Days 1 to Day 8) and 425 mL (about 14.0 oz) during the entire study (from screening to the final visit on Day 11). For comparison, a standard blood donation at a blood collection center, once in a 56-day period, is about 500 mL (2 cups) of blood.

Additional blood samples may be drawn during the study, if the study staff considers it necessary for monitoring your health.

Blood samples and collected data will only be used for this study. Blood samples left after all routine clinical laboratory testing is done will be discarded by the clinical safety laboratory.

#### YOUR ROLE IN THIS STUDY

Taking part in a research study can be an inconvenience to your daily life. Please consider the study time commitments and responsibilities as a research subject when you are deciding to participate. Your responsibilities as a subject include the following:

- You cannot participate in this study if you have participated in a prior study within the past 30 days.
- We ask you to provide accurate responses to questions about your past medical and surgical history (illnesses and surgeries you had including abnormal lab tests, X-rays, and other procedures), medications you are taking, medications you are allergic to and your family history. Failure to respond accurately may result in side-effects that may be harmful after you receive the study drug(s).
- You must read, and agree to follow, the House Rules at the Research Site if you want to
  take part in this study. House Rules discuss proper behavior at the Research Site and are
  important to ensure your safety and make sure the study results are accurate. Failure to
  follow these rules may result in reduced compensation or involuntary discharge from this
  study.
- You must report any side effects and medical problems to the study staff.
- You must give true and complete answers to any questions.
- You must be able to comply with the study procedures and visit schedule.
- You must follow all instructions from the study staff.
- You must inform the study staff if you decide to discontinue your participation in the study. If you decide to discontinue your participation in the study, you may be asked to consent to stay in the study and complete any remaining procedures for the most recent study treatment period. If you do not consent to complete any remaining procedures, you will be asked to complete the early termination visit procedures as described in this consent form.
- You must agree to use an effective method of contraception, as defined later in this consent form, throughout the study and for 30 days after the last dose. If you are male, you must agree not to donate sperm for 30 days after dosing and, if you are sexually active, you and partner to use safe contraception.
- You must not do any strenuous activity for 2 days before the dosing and at any time during the study until discharge on Day 8, and for 24 hours before the out-patient follow up visit on Day 11 (+3 days).
- You must not consume alcohol until your discharge from the clinical site on Day 8 and recommended to avoid alcohol during the out-patient follow-up period until Day 11 (+3 days) (final visit). *Tell the study doctor if you consumed any alcoholic beverages during this time.*
- You must not use marijuana or other illegal drugs during the study.
- You will be advised to avoid smoking after screening. Smoking is prohibited during the in-patient period of the study (Day -1 to Day 8) and recommended to avoid smoking during the follow-up out-patient period to the end of the study (Day 11).
- You must not participate in another research study at any time during this study or continue participating in another study and have blood draws. This includes studies of a drug, biologic (such as vaccine or proteins), device, or blood product.

# PROHIBITED MEDICATIONS, VACCINATIONS, and BLOOD DONATIONS

Additional restrictions to ensure the health and safety of study subjects are listed below:

- You must not take any prescription medications within 14 days before check-in on Day -1 (a day before the start of study drug infusions) or during the study. Certain drugs should be avoided for a longer period before taking the study drug. (See Risks of study drug(s) below).
- You will continue taking birth control medications that you were already using. Certain over-the counter medications may be permitted if approved by the study staff. *Please report all prescription medications you are taking*.
- You must not take any non-prescription medications, herbs, vitamins, or nutritional supplements from the time of screening (about 14 days before dosing) to the end of the study (Day 11), except for single doses of acetaminophen up to 1,000 mg. Certain non-prescription medications are prohibited if taken 14 days before dosing, and others may be permitted if approved by the study staff. *Please report all non-prescription medications*, herbs, vitamins, or nutritional supplements you are taking.
- You must not donate any blood or blood products (red cells, white cells, platelets, plasma) during the course of this study. Tell the study doctor if you donated any blood or blood products within 3 months before dosing. If you did, we could delay your screening.
- You must not receive any blood or blood products during this study unless it is medically necessary.

# RISKS OF STUDY DRUGS

# Observed Risks with ZID:

There were no identified risks associated with ZID in completed human studies in 91 healthy subjects who were given IV single doses ranging from 250 mg to 6 grams daily. The most common side effects, reported by more than one subject, were:

- Headache
- Diarrhea
- Infrequent bowel movements
- Irritation at the injection site

Other side effects that were reported less frequently were:

- Muscle aches
- Numbness around the mouth
- Vaginal discomfort or discharge (in females)

All side effects were mild. ZID was safe and well-tolerated and there were no clinically important changes in laboratory tests and ECGs during that study.

# Potential Risks with ZID:

Until more clinical experience with ZID is available, similar undesirable effects as observed for other drugs should be anticipated. Special attention will be paid to signs and symptoms of allergic reactions. Further testing is needed to understand the potential for ZID to cause mutations and

cancer. Long-term studies in animals and humans are not available. Due to the short duration of study treatment with ZID, the risk of cancer is low.

# Observed risks with ERT:

ERT has been licensed as an antibiotic since 2001 and has been used by patients in the recommended dose (1 gram daily) and by healthy people in research studies at doses (2 gram and 3 gram) that will be used in this study. The most common side effects have been:

- Diarrhea
- Irritation of the infusion vein
- Nausea
- Headache
- Vaginitis (in females)

# Rarely, ERT can cause:

- Diarrhea
- Dizziness
- Increase the risk of seizures, especially in people who have a history of seizures or a condition that makes them more sensitive to seizures.

ERT does not cause changes that increase the risk of cancer.

# **Potential Drug Interactions:**

There are no clinical data on drug interactions with the WCK 6777 (ERT+ZID). However, based on the knowledge about the metabolism of the study drugs and their excretion from the urine, the following drugs should be avoided from 14 days before the first dose to the end of the study:

- Lasix (Furosemide)
- Probenecid
- Other drugs that interact with OTA3 (Adefovir, Anagliptin, Baricitinib, Cefaclor, Cimetidine, Ciprofloxacin (Systemic), Clofarabine, Eluxadoline, Empagliflozin, Ketoprofen, Methotrexate, Mycophenolate, PEMEtrexed, Penicillin G (Parenteral/Aqueous), Penicillin G Benzathine, Penicillin G Procaine, Penicillin V Benzathine, Penicillin V Potassium, Zidovudine).
- Valproic acid

#### Use During Pregnancy and Lactation:

The effects of the study drugs on the pregnant mother and the fetus have not been well studied Therefore, you should not participate in the study if you are pregnant or plan to become pregnant during the study.

ERT has been reported to be detected in maternal milk. Therefore, you should not participate in the study if you are breastfeeding.

# Overdose:

There is no specific antidote in case of overdose. The same measures as recommended for other antibiotics (treatment cessation, adequate hydration, and kidney dialysis) will be provided as medically necessary.

# Drug Abuse and Dependency:

No clinical experience available.

# Potential Risks of WCK 6777 (ERT + ZID):

This is the first time that ERT and ZID are used in people together and there is no information on their side effects; this study will provide some answers.

It is anticipated that the symptoms could be the same as known for each drug separately. Testing before the clinical study did not show any interactions among the two drugs in standard tests of predicting additional side effects of drugs in humans.

#### **BLOOD SAMPLE RISKS**

There may be side effects of drawing blood with a needle and/or IV tubes and IV catheter placement. Local pain, bruising, bleeding, redness, swelling, or induration (palpable hard area) might occur at the site of the needle stick where blood is drawn. Infection at the infusion site or blood draw site is possible but unlikely as aseptic technique will be used. There is a possibility of dizziness or fainting while your blood is being drawn. Precautions will be taken to minimize the above side effects. There is a small risk your blood counts will decrease slightly during the course of the study, but not expected to cause anemia (low blood counts that cause symptoms and need treatment). Any symptoms that may occur are usually reversible with good nutrition and drinking fluids.

#### **ECG RISKS**

ECG patched may case a skin reaction such as redness or itching. You may also experience localized skin discomforts and/or hair loss associated with the placement of ECG patches.

# **UNKNOWN RISKS**

You may have side effects or discomforts that are not listed in this form. Some side effects may not be known yet. New ones could happen to you. Tell the study staff right away if you have any problems.

# **INFORMATION ON BIRTH CONTROL**

#### **Females:**

The effects of study drug(s) on the unborn child are not known at this time. Therefore, it is important that women who are pregnant, may become pregnant or who are breastfeeding NOT participate in this study. If you are a woman who can get pregnant, you <u>must</u> use an acceptable form of birth control that is very effective in preventing pregnancy. You must agree to use birth control for at least 30 days after dosing. You agree to avoid becoming pregnant during this study.

The following are acceptable forms of birth control for this study:

- Progestin implants.
- Intrauterine devices (IUD).
- Surgery to prevent pregnancy in females (such as bilateral tubal ligation, salpingectomy [removal of the tubes], oophorectomy [removal of the ovaries], or hysterectomy [removal of the uterus]).
- Abstinence.

# Tell the study staff if you use any other forms of birth control.

If at any time during this study you think you may be pregnant, you are requested to contact the study doctor at the telephone number listed on the first page of this form.

#### Males:

The effect of study drug(s) on the unborn child is unknown at this time. The effect of the study drug on the male reproductive system is unknown. Therefore, you must agree to use an acceptable form of birth control from dosing with study drug through at least 30 days after the last dose. Acceptable birth control means not having sex (abstinence) or having a vasectomy. If you are sexually active, you should agree to use a condom with spermicide throughout this study and for at least 30 days after dosing. **Tell the study staff if you use any other form of birth control.** 

You should also not donate sperm for 30 days after the last dose.

It is also recommended that you make certain that your female partner is also using an acceptable form of birth control if you have not had a vasectomy and are using a condom. If you think that your partner may be pregnant at any time during this study to 30 days after dosing, you are requested to contact the study doctor at the telephone number listed on the first page of this form.

# **REPORTING PREGNANCY**

If you are a woman, you should report to the study staff if you miss your period and suspect you are pregnant or if you become pregnant during the 30 days after dosing. With your permission, you will continue to be followed for safety during this study. You are requested to provide pregnancy outcome to the study staff upon delivery or pregnancy termination.

If you are a male and your female partner becomes pregnant during the 30 days after dosing, we ask you to inform study staff of the pregnancy and provide pregnancy outcome upon delivery or pregnancy termination.

# INFORMATION ON USE OF ALCOHOL, MARIJUANA OR OTHER ILLEGAL DRUGS

You are not allowed to use alcohol, marijuana or other illegal drugs (such as cocaine, etc.) because they may cause you serious harm and are strictly forbidden while you are in this study. You will be tested for drugs and alcohol at Screening, and on Day -1. If you are found to be in possession of or using marijuana or other illegal drugs at the Research Site, then Altasciences Clinical Kansas, Inc. is obligated to report the use of marijuana or other illegal drugs to the appropriate legal authorities.

# INFORMATION ON ACTIVITIES TO AVOID

You should avoid excessive exercise from at least 2 days before your admission to the Research Site to after the discharge on Day 8 after dosing and 24 hours before your last follow-up visit (Day 11).

# **NEW INFORMATION ABOUT STUDY DRUG(S)**

The study doctor or study staff will discuss with you any important new information, findings or changes to the way the research will be performed that may affect your decision to remain in this study. If this happens, you will be asked to decide if you want to keep taking part in this study. You may be given an additional informed consent and will be asked to agree in writing that you were told about these new findings.

# BENEFITS TO THE STUDY SUBJECT

The goal of this research study is to provide scientific information. You will not receive any medical benefits. This study may help doctors and scientists learn things about the study drug that will help others.

# **ALTERNATE THERAPY**

This is a clinical research study. It is not treatment or therapy. The other choice is to not participate in this study.

# PAYMENT FOR PARTICIPATION

If, after screening, you are enrolled in the study and complete all the study visits, you will receive a total of up to \$4,300.00 at the completion of your participation in the study to help cover the costs of your participation and compensate you for your time. If after enrollment your participation is ended early, or if you withdraw for any reason, the amount you will be paid will be prorated and the payment made when your participation in the study ends. This means that you will receive payment only for the portion of the study that you completed and only after your participation in the study has been completed. Payment will be prorated as follows:

| Visit 1 | Screening | \$150 |
|-------------------|----------------------------------------------|---------|
| Visit 2 | Day -1 Admit | \$375 |
| Visits 3-9 | Days 1 to Day 7 In-house | \$2,625 |
| Visit 10 | Day 8 Discharge | |
| Visit 11 | Day 11 Follow-Up Office Visit / End of Study | \$225 |
| Completion Amount | | \$925 |
| Total | \$4,300 | |

Visit 1 will be compensated in the amount of \$150 at the completion of the visit. Visits 2 through 10 (8 overnight stays) will be compensated in the amount of \$3,000 (\$375 per overnight stay) at discharge on Visit 10.

Visit 11 will be compensated in the amount of \$225 at the completion of the visit.

Compensation will be issued in the form of a check, pre-loaded MasterCard, or cash. The form of compensation will be determined by the study staff.

For any outpatient visit that occurs on a weekend, the associated compensation will be paid on the next business day.

Unscheduled visits may be compensated up to \$50 as determined by the study staff.

All visits must be completed within the scheduled timeframe in order to receive the end of study completion amount of \$925 on Visit 11. Failure to complete all visits within the allowable timeframe will make you ineligible to receive the completion amount.

Money may be deducted from your study compensation if you do not follow the in-house rules or other reasonable instructions given by the study staff. For example, if illegal substances are brought into the research site or you are found to be using an illegal substance while in house, up to half of your previously earned amount may be deducted and you may be withdrawn from the study as determined by the study staff.

If you withdraw or are withdrawn from the study early, you will only be compensated for the visits that you complete.

If you discontinue from the in-house portion of the study early for any reason, you will be compensated one night's earned stipend the same day you discharge from the study.

The remainder of your earned in-house stipend will be compensated to you on the originally scheduled study day/date of discharge from the in-house portion of the study.

You may be required to report the compensation received for this study to the Internal Revenue Service as taxable income. According to the IRS (Internal Revenue Service) guidelines, you will be responsible for paying taxes on any compensation that you receive from your study participation. Altasciences Clinical Kansas, Inc. will send you a 1099-form for this purpose. Altasciences Clinical Kansas, Inc. will also report to the IRS any compensation that you receive that totals \$600.00 or more for the calendar year. You must tell Altasciences Clinical Kansas, Inc. of your new mailing address if you move after your participation in a study. This is to make sure you receive your 1099 for your year-end tax reporting.

# **COMPENSATION FOR INJURY**

• In the event you experience an adverse reaction (side-effect), illness or injury during this study, you should immediately seek treatment. It is important that you tell your study doctor if you have experienced one of these events. You must contact the study staff at the telephone number listed on the first page of this form as soon as you are able. You may obtain medical care in the same way as you would ordinarily receive any other medical treatment. Immediate necessary care, emergency treatment, and professional services will be available to research subjects just as they are to the community generally. No long-term medical care or financial compensation for research-related injuries will be provided by the NIH or the Federal Government.

- Medical care will be given to you at no cost if you are injured because of being in this study.
- While you are in this study, you may be injured because of your personal conduct or during activities, which are not part of this study. There are no plans to pay you for these types of injuries.

### **COSTS TO YOU**

There is no cost to you to participate in this study. You do not have to pay for any study-related medicines, procedures, or study treatment at the Research Site during this study.

# **SOURCE OF FUNDING**

This research study is being funded by NIAID/NIH, which has a contract with a company named DVC to do studies like this one. Altasciences Clinical Kansas, Inc. has signed a contract with IQVIA, Inc., a subcontractor of DVC, to conduct this research study under the direction of Martin Kankam, MD.

# **VOLUNTARY PARTICIPATION IN THIS STUDY**

Your participation in this study is voluntary. You will be starting this study of your own free will and without any kind of pressure. You may quit this study any time you wish. If you withdraw from this study, you will not be penalized. You will not lose any benefits to which you were otherwise entitled.

If you have health problems, you will get medical attention. You may be withdrawn from this study by the study staff and/or the sponsor of this study, without your consent, if it is in your best medical interest. It is possible that the study staff and/or sponsor may think you can stay in this study. You must decide what you want to do.

The study staff may stop your participation in this study at any time without your consent for any of the following reasons:

- If you don't follow the study staff's instructions;
- Something serious happens to you which may require treatment;
- The study staff decides it is in the best interest of your health, and welfare to discontinue further participation;
- You do not later consent to any future changes that may be made in the study plan.

The sponsor may stop this study for other reasons not known now.

The FDA or the Institutional Review Board (IRB, see below) may also terminate this study if there are safety concerns.

#### IF YOU WITHDRAW FROM THE STUDY

If you do not complete this study for any reason, you will be asked to undergo a physical exam, vital signs measurement, 12-lead ECG, blood and urine laboratory tests, and tests for the measurement of study drug concentration in your blood if early termination occurs within 24

hours of dosing. This is needed to identify any changes that may have occurred after you began to take the study drug and to protect your safety, health, and welfare.

If you received any amount of the study drug but withdraw from the trial within 24 hours after dosing, you will be encouraged to continue follow-up (with your consent) for safety assessments. We may also ask you to provide PK blood and urine sample(s) to complete scheduled collection if you had received study drug on the day you withdrew from the study.

#### CERTIFICATE OF CONFIDENTIALITY

To help us protect your privacy, we have a Certificate of Confidentiality from NIH. The study staff can use this Certificate to legally refuse to give information that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings, for example, if there is a court subpoena. The study staff will use the Certificate to resist any demands for information that would identify you, except for reporting of communicable diseases, such as Hepatitis Virus and HIV infections, to state and local health departments, or for reporting possession or use of marijuana or other illegal drugs while at the Research Site to the appropriate legal authorities.

A Certificate of Confidentiality does not prevent disclosure of your information to the NIH, FDA, or federal funding agency. Information from this study will be given to DMID and Wockhardt Ltd., the pharmaceutical organization developing WCK 6777 and other drugs for the treatment of infectious diseases. Any persons or companies, which are contracted by the sponsor for conducting this study, measuring drug level in blood samples, monitoring the execution of this study, and analyzing the data, will have access to the research information during and after this study, The information will also be given to the FDA. It may be given to governmental agencies in other countries where the study drug may be considered for approval.

Medical records which identify you and the consent form signed by you will be looked at and/or copied for research or regulatory purposes by:

- The sponsor
- An agent for the sponsor
- An agent for the study doctor
- The FDA
- Department of Health and Human Services (DHHS) agencies
- The Institutional Review Board, Advarra IRB.

Absolute confidentiality cannot be guaranteed because of the need to give information to these parties. The results of this research study may be presented at meetings or in publications. Your identity will not be disclosed in those presentations.

- Altasciences Clinical Kansas, Inc. will handle the medical information obtained in this study with the strictest confidence. It will be protected as required by laws and/or regulations. It will not be made publicly available.
- If the results of this study are published, you will not be identified by name.
- Your identity will not be disclosed to anyone else, unless required by law.

By signing this consent, you authorize Altasciences Clinical Kansas, Inc. to verify your study participation history with other businesses that conduct clinical research studies.

A Certificate of Confidentiality does not prevent you or a member of your family from voluntarily releasing information about yourself or your involvement in this research. If you give your consent to release information to a medical care provider, an insurer, or other person to receive research information, then the researchers will not withhold that information.

#### PRIMARY CARE PHYSICIAN NOTIFICATION

We would like your permission to contact the doctor you see regularly to let them know that you are taking part in this study. It is important for all your doctors to know that you may be taking an experimental drug. Your doctor will want to know and think about all the drugs you are taking before giving you any new ones. While you are in the study, the study doctor will ask about your symptoms. If you have symptoms after the study ends, your other doctor may want to contact the study personnel.

If you agree, your primary care physician (regular doctor) will be informed of your participation in the study. Indicate your choice below by initialing only one (1) section below.

| Initials | I do not have a primary care physician. |
|---|---|
| Initials | I do not want my primary care physician notified. |
| Initials | I would like my primary care physician notified and below is my physician's contact information. Physician's Name: Address: Phone No.: |

# WHOM TO CONTACT ABOUT THIS STUDY

During the study, if you experience any medical problems, suffer a research-related injury, or have questions, concerns, or complaints about the study, such as:

- Whom to contact in the case of a research-related injury or illness;
- Payment or compensation for being in the study, if any;
- Your responsibilities as a research subject;
- Eligibility to participate in the study;

- The study doctor's or study site's decision to withdraw you from participation;
- Results of tests and/or procedures;

# <u>Please contact the study doctor at the telephone number listed on the first page of this consent document.</u>

If you seek emergency care, or hospitalization is required, alert the treating physician that you are participating in this research study.

An institutional review board (IRB) is an independent committee established to help protect the rights of research subjects. If you have any questions about your rights as a research subject, and/or concerns or complaints regarding this research study, contact:

By mail: Study Subject Adviser

Advarra IRB

6100 Merriweather Dr., Suite 600

Columbia, MD 21044

or call toll free: 877-992-4724

• or by email: adviser@advarra.com

Please reference the following number when contacting the Study Subject Adviser: <u>Pro00066629</u>

# **CONSENT and AUTHORIZATION**

I have read all information in this document, and all my questions have been answered to my satisfaction. I voluntarily consent to participate in this study. I will be given a signed and dated copy of this consent form, and have been told the description of the study drug, and the name, address and phone number of the study doctor. My signature gives my consent to participate. I authorize the release of my medical records and health information related to this study, including my signed and dated consent form and any addendum, to the sponsor and its representatives, the FDA, Advarra IRB and other regulatory agencies as described above. By signing and dating this form, I have not given up any of my legal rights as a research subject.

| Print Subject's Name | Date |
|------------------------------------------------|------|
| Subject's Signature | |
| Person Obtaining Informed Consent Printed Name | |
| Person Obtaining Informed Consent Signature | Date |
| Witness Printed Name | |
| Witness Signature | Date |
| Investigator's Signature* | Date |

<sup>\*</sup>The Investigator's signature evidences only that the Investigator has reviewed the consent form and the signatures of the subject, person obtaining consent, and witness, for compliance.